CLINICAL TRIAL: NCT03389711
Title: INCMNSZ Early Rheumatoid Arthritis Cohort
Brief Title: INCMNSZ - Rheumatoid Arthritis Cohort
Acronym: IRAC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Institute of Medical Sciences and Nutrition, Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Virginia Pascual Ramos, Lead Investigator of the Rheumatoid Arthritis Clinic, National Institute of Medical Sciences and Nutrition, Salvador Zubiran
Other Study IDs: IRE-274-10/11-1
Record Dates: First submitted 2017-12-14; First posted 2018-01-04 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2021-08

CONDITIONS: Early Rheumatoid Arthritis; Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis Mexico; Early Rheumatoid Arthritis Cohort Mexico
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples to asses serological status (rheumatoid arthritis antibodies)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Combination Product: DMARD´s and multidisciplinary treatment — At study enrollment, medical history, disease-specific autoantibodies, ACR 1987 classification criteria for RA were applied. Medical evaluations were standardized and included at least 66 swollen and 68 tender joint counts, acute reactant-phase determinations , patient and physician reported outcomes, comorbidity established by record review, and treatment assessments (name, dose and schedule of all drug they were taking) along with an evaluation of persistence, at six-month intervals.
  Patients were evaluated by a single rheumatologist every two months during the first two years of follow-up, and every two, four or six months thereafter.
  Also the following scores: Michigan Hand Outcome Questionnaire (MHQ), Disabilities of the Arm, Shoulder and Hand Outcome Measure (DASH),Mayor Depressive Episodes (MDE) was defined using the Mini International Neuropsychiatric Interview and the severity of depressive symptoms was assessed with the Beck Depression Inventory (BDI-II).

SUMMARY:
Identify Rheumatoid Arthritis patients diagnose within first 12 months since the beginning of the disease related symptoms. Initiate proper treatment according to international standards in order to achieve remission/low disease activity status.

DETAILED DESCRIPTION:
* Provide an standardized follow up by a multidisciplinary specialized team.
* Create a biological (blood) bank to develop future research projects.
* Create a database with the clinical, serologic, radiographic and functional status patients data.
* Define comorbidities and mortality causes.
* Begin an educational program to improve patient disease self-knowledge

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years old
* Fulfilled ACR 1987 classification criteria for RA
* Disease evolution of <1 year when first evaluated, and no specific rheumatic diagnosis except for RA.

Exclusion Criteria:

* Patients with another rheumatic disease, except Sjögren syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán (INCMNSZ) belongs to the National Institutes of Health of México. Patients enrolled in the Early arthritis cohort had a disease duration of <1 year when first evaluated, and no specific rheumatic diagnosis except for RA. Patients had partial health coverage and paid for their physician's consultations, laboratory investigations and for their treatment that was prescribed by the rheumatologist in charge of the clinic, and was "treat to target" oriented.
Sampling Method: Non-Probability Sample
Enrollment: 237 (Estimated)
Dates: Start 2004-02-04 (Actual); Primary Completion 2024-02-04 (Estimated); Study Completion 2024-02-04 (Estimated)

PRIMARY OUTCOMES:
Disease activity status | During the first two years of follow up: the evaluations will be every 2 months. After those years: the evaluations will be every 2, 4 or 6 months depending on disease activity status.
  Describe the disease activity score using DAS 28 ESR

SECONDARY OUTCOMES:
Change from Baseline of the Patient Reported Outcome : HAQ (Health Assessment Questionnarie) | During the first two years of follow up: the evaluations will be every 2 months. After those years: the evaluations will be every 2, 4 or 6 months depending on disease activity status.
  To describe the changes in every visit in the HAQ score
Change from Baseline of the Patient Reported Outcome: RADAI (Rheumatoid Arthritis Disease Activity Index) | During the first two years of follow up: the evaluations will be every 2 months. After those years: the evaluations will be every 2, 4 or 6 months depending on disease activity status.
  To describe the changes in every visit in the RADAI score
Change from Baseline of the Patient Reported Outcome : SF-36 (Short Form Health Survey) | During the first two years of follow up: the evaluations will be every 2 months. After those years: the evaluations will be every 2, 4 or 6 months depending on disease activity status.
  To describe the changes in every visit in the SF-36 score
Predictors of health care drop-out | During the first two years of follow up: the evaluations will be every 2 months. After those years: the evaluations will be every 2, 4 or 6 months depending on disease activity status.
  Identify and describe patients from an inception ongoing cohort with recent onset RA at inclusion, who dropped out of health care during their follow-up
Mayor Depressive Episodes (MDE) | During the first two years of follow up: the evaluations will be every 2 months. After those years: the evaluations will be every 2, 4 or 6 months depending on disease activity status.
  Investigate associations between major depressive episodes (MDE), concordance with therapy (CwT) and disease outcomes in rheumatoid arthritis patients.
Michigan Hand Outcome Questionnarie (MHQ | During the first two years of follow up: the evaluations will be every 2 months. After those years: the evaluations will be every 2, 4 or 6 months depending on disease activity status.
  To assess a variety of hand and upper extremity injuries related to Rheumatoid Arthritis
Disabilities of the Arm, Shoulder and Hand Outcome Measure (DASH) | During the first two years of follow up: the evaluations will be every 2 months. After those years: the evaluations will be every 2, 4 or 6 months depending on disease activity status.
  To measure upper-extremity disability and symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Pascual, MD, Principal Investigator — INCMNSZ
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City, Tlalpan, Mexico

IPD SHARING:
Plan to Share IPD: No
It is undecided yet.

REFERENCES:
- [Result] Contreras-Yanez I, Pascual-Ramos V. Predictors of health care drop-out in an inception cohort of patients with early onset rheumatoid arthritis. BMC Musculoskelet Disord. 2017 Jul 28;18(1):321. doi: 10.1186/s12891-017-1670-6. PMID 28754110
- [Result] Contreras-Yanez I, Guaracha-Basanez G, Ruiz-Dominguez D, Pascual-Ramos V. Patient's perspective of sustained remission in rheumatoid arthritis. BMC Musculoskelet Disord. 2017 Sep 2;18(1):379. doi: 10.1186/s12891-017-1717-8. PMID 28865423
- [Result] Romero-Guzman AK, Menchaca-Tapia VM, Contreras-Yanez I, Pascual-Ramos V. Patient and physician perspectives of hand function in a cohort of rheumatoid arthritis patients: the impact of disease activity. BMC Musculoskelet Disord. 2016 Sep 15;17:392. doi: 10.1186/s12891-016-1246-x. PMID 27628666
- [Result] Atisha-Fregoso Y, Lima G, Pascual-Ramos V, Banos-Pelaez M, Fragoso-Loyo H, Jakez-Ocampo J, Contreras-Yanez I, Llorente L. Rheumatoid Arthritis Disease Activity Is Determinant for ABCB1 and ABCG2 Drug-Efflux Transporters Function. PLoS One. 2016 Jul 21;11(7):e0159556. doi: 10.1371/journal.pone.0159556. eCollection 2016. PMID 27442114
- [Result] Contreras-Yanez I, Pascual-Ramos V. Window of opportunity to achieve major outcomes in early rheumatoid arthritis patients: how persistence with therapy matters. Arthritis Res Ther. 2015 Jul 11;17(1):177. doi: 10.1186/s13075-015-0697-z. PMID 26162892
- [Result] Galicia-Hernandez G, Parra-Salcedo F, Ugarte-Martinez P, Contreras-Yanez I, Ponce-de-Leon A, Pascual-Ramos V. Sustained moderate-to-high disease activity and higher Charlson score are predictors of incidental serious infection events in RA patients treated with conventional disease-modifying anti-rheumatic drugs: a cohort study in the treat-to-target era. Clin Exp Rheumatol. 2016 Mar-Apr;34(2):261-9. Epub 2016 Mar 3. PMID 26939612
- [Result] Parra-Salcedo F, Contreras-Yanez I, Elias-Lopez D, Aguilar-Salinas CA, Pascual-Ramos V. Prevalence, incidence and characteristics of the metabolic syndrome (MetS) in a cohort of Mexican Mestizo early rheumatoid arthritis patients treated with conventional disease modifying anti-rheumatic drugs: the complex relationship between MetS and disease activity. Arthritis Res Ther. 2015 Feb 20;17(1):34. doi: 10.1186/s13075-015-0549-x. PMID 25889060
- [Result] Cabrera-Marroquin R, Contreras-Yanez I, Alcocer-Castillejos N, Pascual-Ramos V. Major depressive episodes are associated with poor concordance with therapy in rheumatoid arthritis patients: the impact on disease outcomes. Clin Exp Rheumatol. 2014 Nov-Dec;32(6):904-13. Epub 2014 Sep 5. PMID 25190569
- [Result] Sanchez T, Contreras-Yanez I, Elias-Lopez D, Aguilar Salinas CA, Pascual-Ramos V. Prevalence of lipid phenotypes, serum lipid behaviour over follow-up and predictors of serum lipid levels in a cohort of Mexican Mestizo early rheumatoid arthritis patients treated with conventional disease-modifying anti-rheumatic drugs. Clin Exp Rheumatol. 2014 Jul-Aug;32(4):509-15. Epub 2014 Jul 8. PMID 25005131
- [Result] Pascual-Ramos V, Contreras-Yanez I, Rivera-Hoyos P, Enriquez L, Ramirez-Anguiano J. Cumulative disease activity predicts incidental hearing impairment in patients with rheumatoid arthritis (RA). Clin Rheumatol. 2014 Mar;33(3):315-21. doi: 10.1007/s10067-014-2485-6. Epub 2014 Jan 18. PMID 24435352
- [Result] Pascual-Ramos V, Contreras-Yanez I. Motivations for inadequate persistence with disease modifying anti-rheumatic drugs in early rheumatoid arthritis: the patient's perspective. BMC Musculoskelet Disord. 2013 Dec 1;14:336. doi: 10.1186/1471-2474-14-336. PMID 24289729
- [Result] Contreras-Yanez I, Rull-Gabayet M, Vazquez-Lamadrid J, Pascual-Ramos V. Radiographic outcome in Hispanic early rheumatoid arthritis patients treated with conventional disease modifying anti-rheumatic drugs. Eur J Radiol. 2011 Aug;79(2):e52-7. doi: 10.1016/j.ejrad.2011.03.036. Epub 2011 Apr 8. PMID 21477956
- [Result] Contreras-Yanez I, Ponce De Leon S, Cabiedes J, Rull-Gabayet M, Pascual-Ramos V. Inadequate therapy behavior is associated to disease flares in patients with rheumatoid arthritis who have achieved remission with disease-modifying antirheumatic drugs. Am J Med Sci. 2010 Oct;340(4):282-90. doi: 10.1097/MAJ.0b013e3181e8bcb0. PMID 20881757
- [Result] Pascual-Ramos V, Contreras-Yanez I, Cabiedes-Contreras J, Rull-Gabayet M, Villa AR, Vazquez-Lamadrid J, Mendoza-Ruiz JJ. Hypervascular synovitis and American College of Rheumatology Classification Criteria as predictors of radiographic damage in early rheumatoid arthritis. Ultrasound Q. 2009 Mar;25(1):31-8. doi: 10.1097/RUQ.0b013e3181981df0. PMID 19276959
- [Result] Pascual-Ramos V, Contreras-Yanez I, Villa AR, Cabiedes J, Rull-Gabayet M. Medication persistence over 2 years of follow-up in a cohort of early rheumatoid arthritis patients: associated factors and relationship with disease activity and with disability. Arthritis Res Ther. 2009;11(1):R26. doi: 10.1186/ar2620. Epub 2009 Feb 19. PMID 19228421